CLINICAL TRIAL: NCT02149524
Title: A Phase III Randomised, Double-Blind, Parallel Group, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity Between SB3 (Proposed Trastuzumab Biosimilar) and Herceptin® in Women With Newly Diagnosed HER2 Positive Early or Locally Advanced Breast Cancer in Neoadjuvant Setting
Brief Title: A Study to Compare the Effect of SB3 and Herceptin® in Women With HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB3-G31-BC; 2013-004172-35 (EudraCT Number)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-03

CONDITIONS: HER2 Positive Early or Locally Advanced Breast Cancer
Keywords: HER2 Positive Breast Cancer; Trastuzumab; Biosimilar
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herceptin (trastuzumab) (Active Comparator): Intravenous administration
  Interventions: Drug: Herceptin (trastuzuamb)
- SB3 (proposed trastuzumab biosimilar) (Experimental): Intravenous administration
  Interventions: Drug: SB3 (proposed trastuzumab biosimilar)

INTERVENTIONS:
Drug: Herceptin (trastuzuamb) — Intravenous administration
  Other Names: Herceptin
  Arms: Herceptin (trastuzumab)
Drug: SB3 (proposed trastuzumab biosimilar) — Intravenous administration
  Arms: SB3 (proposed trastuzumab biosimilar)

SUMMARY:
A Phase III Randomised, Double-Blind, Parallel Group, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity between SB3 (proposed trastuzumab biosimilar) and Herceptin® in Women with Newly Diagnosed HER2 Positive Early or Locally Advanced Breast Cancer in Neoadjuvant Setting

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-65 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Non-metastatic, unilateral newly diagnosed primary breast cancer of clinical stage II to III including inflammatory breast cancer with:

  1. tumour size ≥ 2 cm
  2. histologically confirmed primary invasive carcinoma of the breast
  3. HER2-positivity confirmed by a central laboratory or an accredited local laboratory and defined as immunohistochemistry (IHC) 3+ or fluorescence in situ hybridisation (FISH)+
* Known hormone receptor (oestrogen receptor and progesterone receptor) status
* Baseline left ventricular ejection fraction (LVEF) ≥ 55% measured by echocardiography or multiple gated acquisition (MUGA) scan
* Subjects must be able to provide informed consent, which must be obtained prior to any study related procedures

Exclusion Criteria:

* Metastatic (stage IV) or bilateral or multifocal/multicentric breast cancer
* History of any prior invasive breast carcinoma, except for subjects with a past history of ductal carcinoma in situ (DCIS) and/or lobular carcinoma in situ (LCIS) treated with surgery only
* Past or current history of malignant neoplasms within 5 years prior to Randomisation, except for curatively treated carcinoma in situ of uterine cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin (malignant neoplasms occurring more than 5 years prior to Randomisation are permitted if curatively treated with surgery only)
* Previous history of radiation therapy, immunotherapy, chemotherapy or biotherapy (including prior HER2 directed therapy) Major surgery within 4 weeks prior to Randomisation and minor surgery within 2 weeks prior to Randomisation (major surgery is defined as surgery which requires general anaesthesia)
* Serious cardiac illness that would preclude the use of trastuzumab such as:

  1. history of documented congestive heart failure (CHF) (New York Heart Association, NYHA, class II or greater heart disease)
  2. LVEF < 55% by echocardiography or MUGA scan
  3. angina pectoris requiring anti-anginal medication
  4. evidence of transmural infarction on electrocardiogram (ECG)
  5. uncontrolled hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg)
  6. clinically significant valvular heart disease
  7. high risk uncontrolled arrhythmias
* Serious pulmonary illness enough to cause dyspnoea at rest or requiring supplementary oxygen therapy
* Known history of hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection
* Other concurrent serious illnesses that may interfere with planned therapy including severe cardiovascular, pulmonary, metabolic or infectious conditions
* Known hypersensitivity to the investigational product (IPs), non-IPs or any of the ingredients or excipients of the IPs or non-IPs
* Known hypersensitivity to murine proteins
* Known history of dihydropyrimidine dehydrogenase (DPD) deficiency
* Pre-existing peripheral sensory or motor neuropathy ≥ grade 2, defined by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0
* Pregnant or lactating women. A pregnancy test result is required for all women of childbearing potential including women who had menopause onset within 2 years prior to Randomisation. Women of childbearing potential must agree to use contraceptive methods (see section 7.4.2) during the study and 6 months after the last dose of IP
* Concurrent hormonal therapy including birth control pills, ovarian hormone replacement for menopause, selective oestrogen receptor modulator (SERM) either for osteoporosis or breast cancer prevention
* Subjects unwilling to follow the study requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Pivot, Principal Investigator — CHU Besançon Hopital Jean Minjoz Service d'Oncologie Medicale
Locations (1):
- Investigational Site, Prague, Czechia

REFERENCES:
- [Derived] Pivot X, Bondarenko I, Nowecki Z, Dvorkin M, Trishkina E, Ahn JH, Im SA, Sarosiek T, Chatterjee S, Wojtukiewicz MZ, Shparyk Y, Moiseyenko V, Bello M 3rd, Semiglazov V, Lee Y, Lim J. A phase III study comparing SB3 (a proposed trastuzumab biosimilar) and trastuzumab reference product in HER2-positive early breast cancer treated with neoadjuvant-adjuvant treatment: Final safety, immunogenicity and survival results. Eur J Cancer. 2018 Apr;93:19-27. doi: 10.1016/j.ejca.2018.01.072. Epub 2018 Feb 12. PMID 29448072
- [Derived] Pivot X, Bondarenko I, Nowecki Z, Dvorkin M, Trishkina E, Ahn JH, Vinnyk Y, Im SA, Sarosiek T, Chatterjee S, Wojtukiewicz MZ, Moiseyenko V, Shparyk Y, Bello M 3rd, Semiglazov V, Song S, Lim J. Phase III, Randomized, Double-Blind Study Comparing the Efficacy, Safety, and Immunogenicity of SB3 (Trastuzumab Biosimilar) and Reference Trastuzumab in Patients Treated With Neoadjuvant Therapy for Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer. J Clin Oncol. 2018 Apr 1;36(10):968-974. doi: 10.1200/JCO.2017.74.0126. Epub 2018 Jan 26. PMID 29373094

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Started | 438 | 437
Completed | 384 | 380
Not Completed | 54 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar) | Total
Number analyzed (Participants) | 438 | 437 | 875
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data for one subject is missing.
  years
    number analyzed (Participants) | 437 | 437 | 874
    (all) | 49.6 (9.38) | 49.5 (9.51) | 49.6 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 438 | 437 | 875
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Pathologic Complete Response (pCR) Rate of the Primary Breast Tumour
Time Frame: Week 24
Population: Per-protocol set
Measure: Number; unit: percentage of responders
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 398 | 402
percentage of responders | 42.0 | 51.7

2. Secondary Outcome: Total Pathological Complete Response (tpCR) Rate
Time Frame: Week 24
Population: Per-protocol set
Measure: Number; unit: percentage of responders
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 380 | 382
percentage of responders | 35.8 | 45.8

3. Secondary Outcome: Overall Clinical Response Rate (ORR)
Time Frame: Week 24
Population: Per-protocol set
Measure: Number; unit: percentage of responders
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 374 | 383
percentage of responders | 91.2 | 96.3

4. Secondary Outcome: Event-free Survival (EFS)
Time Frame: 1 month after last dose of investigational product
Population: Per-protocol set
Measure: Number; unit: percentage of subjects without event
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 398 | 402
percentage of subjects without event | 92.7 | 93.8

5. Secondary Outcome: Overall Survival (OS)
Time Frame: 1 month after the last administration of investigational product
Population: Per-protocol set
Measure: Number; unit: percentage of subjects alive
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
Number analyzed (Participants) | 398 | 402
percentage of subjects alive | 99.5 | 100.0

ADVERSE EVENTS:
Arm/Group | Herceptin (Trastuzumab) | SB3 (Proposed Trastuzumab Biosimilar)
All-Cause Mortality (participants affected / at risk) | 5/438 | 1/437
Serious Adverse Events (participants affected / at risk) | 58/438 | 56/437
Other Adverse Events (participants affected / at risk) | 420/438 | 426/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Herceptin (Trastuzumab) (N=438) | SB3 (Proposed Trastuzumab Biosimilar) (N=437)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (14) | 10 (11)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Intraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radiation mucositis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (7) | 8 (20)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Herceptin (Trastuzumab) (N=438) | SB3 (Proposed Trastuzumab Biosimilar) (N=437)
Neutropenia (Blood and lymphatic system disorders) | 280 (634) | 293 (654)
Leukopenia (Blood and lymphatic system disorders) | 113 (237) | 125 (259)
Anaemia (Blood and lymphatic system disorders) | 95 (198) | 96 (180)
Nausea (Gastrointestinal disorders) | 135 (388) | 143 (362)
Diarrhoea (Gastrointestinal disorders) | 65 (90) | 91 (143)
Vomiting (Gastrointestinal disorders) | 50 (87) | 61 (110)
Stomatitis (Gastrointestinal disorders) | 51 (88) | 61 (107)
Dyspepsia (Gastrointestinal disorders) | 22 (27) | 26 (39)
Fatigue (General disorders) | 79 (182) | 88 (186)
Asthenia (General disorders) | 55 (162) | 57 (145)
Pyrexia (General disorders) | 37 (48) | 39 (50)
Oedema peripheral (General disorders) | 31 (34) | 18 (27)
Upper respiratory tract infection (Infections and infestations) | 40 (64) | 44 (66)
Radiation skin injury (Injury, poisoning and procedural complications) | 38 (47) | 48 (48)
Procedural pain (Injury, poisoning and procedural complications) | 53 (54) | 39 (41)
Infusion related reaction (Injury, poisoning and procedural complications) | 42 (62) | 37 (53)
Postoperative wound complication (Injury, poisoning and procedural complications) | 21 (21) | 27 (27)
Alanine aminotransferase increased (Investigations) | 83 (150) | 84 (150)
Aspartate aminotransferase increased (Investigations) | 63 (110) | 68 (102)
Neutrophil count decreased (Investigations) | 53 (162) | 53 (124)
White blood cell count decreased (Investigations) | 32 (71) | 25 (69)
Blood alkaline phosphatase increased (Investigations) | 29 (43) | 22 (40)
Decreased appetite (Metabolism and nutrition disorders) | 41 (103) | 40 (78)
Myalgia (Musculoskeletal and connective tissue disorders) | 66 (138) | 63 (148)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (70) | 48 (74)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 20 (21) | 27 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 24 (39) | 23 (39)
Headache (Nervous system disorders) | 32 (51) | 31 (55)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (40) | 30 (42)
Neuropathy peripheral (Nervous system disorders) | 12 (12) | 22 (24)
Insomnia (Psychiatric disorders) | 22 (31) | 22 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (34) | 41 (46)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 25 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 283 (324) | 299 (349)
Rash (Skin and subcutaneous tissue disorders) | 45 (62) | 47 (61)
Nail disorder (Skin and subcutaneous tissue disorders) | 23 (23) | 22 (23)
Lymphorrhoea (Vascular disorders) | 30 (51) | 32 (58)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow Sponsor sixty (60) days to review and comment on them.